CLINICAL TRIAL: NCT02683031
Title: A Prospective Randomized Controlled Trial Investigating Embryonic Development and Clinical Outcome After Using Ca2+ Ionophore in Cases With Previous Fertilization Arrest
Brief Title: Effect of Ca2+ Ionophore on Embryonic Development and Clinical Outcome in Cases With Previous Fertilization Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TopLab Company for ART Laboratories Consultation and Training (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Yasmin Magdi, Senior clinical embryologist, Dar AlMaraa Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #0010010
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Fertilization Arrest
Keywords: fertilization arrest; Cleavage failure; Embryonic development; Calcium ionophore

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Ca2+ ionophore (No Intervention): Patients with previous incomplete ICSI cycle due to fertilization arrest were counseled to underwent a subsequent conventional ICSI cycle.
- With Ca2+ ionophore (Experimental): Patients with previous incomplete ICSI cycle due to fertilization arrest were counseled to underwent a subsequent ICSI cycle combined with artificial oocyte activation using Ca2+ ionophore.
  Interventions: Other: Ca2+ ionophore

INTERVENTIONS:
Other: Ca2+ ionophore — Ca2+ ionophore is a chemical agent used to perform oocyte activation after ICSI. It showed effective treatment to get better fertilization, pregnancy, and healthy livebirth in cases with total or partial fertilization failure.
  Other Names: A23187 Ca2+ ionophore
  Arms: With Ca2+ ionophore

SUMMARY:
We aimed to investigate the efficiency of chemical oocyte activation using readymade Ca2+ ionophore on cases with previously cancelled cases due to fertilization arrest at pronuclear stage i.e: cleavage failure to find out if there is any improvement in embryonic developmental stages.

DETAILED DESCRIPTION:
Many studies reported that Ca2+ ionophore has a positive effect on embryo development in cases with complete or partial fertilization failure. However, only one preliminary report suggested a beneficial effect of Ca2+ ionophore activation in four cases with fertilization arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous history of complete fertilization arrest.
* ovarian stimulation with the GnRH agonist and recombinant FSH in a long protocol.

Exclusion Criteria:

* Female age >40 years

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Blastocyst formation rate | 5 to 7days post oocyte retrival
  Defined as the total number of blastocyst / total number of cleaved Embryos

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Magdi, M.Sc, Principal Investigator — Dar Almaraa fertility and gynacology center; Mona M. Awady, MD, Study Chair — Department of Community Medicine, Faculty of Medicine, Benha University, Benha, Egypt
Locations (1):
- Ahmed el-Damen, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ebner T, Koster M, Shebl O, Moser M, Van der Ven H, Tews G, Montag M. Application of a ready-to-use calcium ionophore increases rates of fertilization and pregnancy in severe male factor infertility. Fertil Steril. 2012 Dec;98(6):1432-7. doi: 10.1016/j.fertnstert.2012.07.1134. Epub 2012 Aug 24. PMID 22921909
- [Background] Ebner T, Montag M; Oocyte Activation Study Group; Montag M, Van der Ven K, Van der Ven H, Ebner T, Shebl O, Oppelt P, Hirchenhain J, Krussel J, Maxrath B, Gnoth C, Friol K, Tigges J, Wunsch E, Luckhaus J, Beerkotte A, Weiss D, Grunwald K, Struller D, Etien C. Live birth after artificial oocyte activation using a ready-to-use ionophore: a prospective multicentre study. Reprod Biomed Online. 2015 Apr;30(4):359-65. doi: 10.1016/j.rbmo.2014.11.012. Epub 2014 Dec 9. PMID 25596904
- [Result] Darwish E, Magdi Y. A preliminary report of successful cleavage after calcium ionophore activation at ICSI in cases with previous arrest at the pronuclear stage. Reprod Biomed Online. 2015 Dec;31(6):799-804. doi: 10.1016/j.rbmo.2015.08.012. Epub 2015 Aug 28. PMID 26507280